CLINICAL TRIAL: NCT02222181
Title: Impact of Pharmacotherapy Management in Patients With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Fernanda Mariana de Oliveira, Master's degree student, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 24947914.5.0000.5426
Record Dates: First submitted 2014-08-04; First posted 2014-08-21 (Estimated); Results first posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-04

CONDITIONS: Alzheimer's Disease
Keywords: elderly, medication adherence,pharmaceutical care
MeSH Terms: conditions — Alzheimer Disease; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacotherapy follow-up (Experimental): patients with Alzheimer's disease
  Interventions: Other: Pharmacotherapy Management

INTERVENTIONS:
Other: Pharmacotherapy Management — * assessment of patient characteristics as alcoholic, smoker, food, drugs
  * Pharmacotherapy follow-up
  * to evaluated medication adherence
  * Assessment of the individual clinical parameters each patient at baseline and after the educational or pharmacy intervention.

SUMMARY:
In Brazil, patients with Alzheimer's disease (AD) receiving free drugs of government. Even having access to, little is known about the effectiveness, safety and adherence of drug therapy in this group of patients. The research aims to promote adherence and develop strategies to address Drug-Related Problems (DRP's) in AD patients elderly of reference centre for the Elderly of Araraquara. The clinical parameters will be assessed at the beginning and after the educational intervention period from April 2014 to April 2015.

DETAILED DESCRIPTION:
Dementia is characterized by memory loss associated with cognitive impairment, which directly interferes in learning process, social and professional performance, besides being the main cause of dementia or Alzheimer's disease (AD). In Brazil, patients are medicated for AD through "Programa de Medicamentos Excepcionais" (Exceptional Drug Program) that ensure the patient´s treatment by providing high cost medications. Even having access to, little is known about the effectiveness, safety and adherence of drug therapy in this group of patients. The research aims to promote adherence and develop strategies to address Drug-Related Problems (DRP's) in AD patients. For this end, we intend to conduct a descriptive, almost experimental and longitudinal uncontrolled research, from April 2014 to December 2015, at the CRIA: "Centro de Referência do Idoso de Araraquara" (Reference Centre for the Elderly of Araraquara). Patients included in the research must have a diagnosis of AD and must be using drugs supplied by the "Programa de Medicamentos Excepcionais". For data collection pharmaceutical care will be employed as a technique, carried out through pharmaceutical meetings, including the steps of initial assessment, care plan (pharmaceutical intervention) and results evaluation. The results will be monitored for pharmacotherapy adherence, cognitive assessment and other clinical parameters related to their health problems and resolution of DRP's before and after the proposed follow-up.The expected outcomes include knowledge of the medication experiences of AD patients, how they influence the adherence and other DRP's and how they can contribute by solving these problems, in addition to the impact evaluation of pharmaceutical care in cognitive improving and other clinical parameters monitored and evaluated individually.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients who are assisted in CRIA, diagnosed with Alzheimer's in use of rivastigmine or donepezil or galantamine, assisted by the "Program for special drugs".
* Be resident in the city of Araraquara / SP
* Accept part of pharmacotherapeutic follow-up;
* Sign the Statement of Informed Consent Form (ICF).

Exclusion Criteria:

* Fold over pharmacotherapy follow-up;
* Being institutionalized;
* Patients unable to respond to collection instruments MMSE and CDR data;
* Patient without phone contact.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda M Oliveira, student, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Centro de Referência do Idoso de Araraquara - CRIA, Araraquara, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strand LM, Cipolle RJ, Morley PC. Documenting the clinical pharmacist's activities: back to basics. Drug Intell Clin Pharm. 1988 Jan;22(1):63-7. doi: 10.1177/106002808802200116. PMID 3349924
- [Background] Arlt S, Lindner R, Rosler A, von Renteln-Kruse W. Adherence to medication in patients with dementia: predictors and strategies for improvement. Drugs Aging. 2008;25(12):1033-47. doi: 10.2165/0002512-200825120-00005. PMID 19021302
- [Background] Lanctot KL, Herrmann N, Yau KK, Khan LR, Liu BA, LouLou MM, Einarson TR. Efficacy and safety of cholinesterase inhibitors in Alzheimer's disease: a meta-analysis. CMAJ. 2003 Sep 16;169(6):557-64. PMID 12975222

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Experimental, longitudinal and non-randomized study, carried out at Centro de Referência do Idoso de Araraquara (CRIA), from 2014 april to 2015 april, with patients in treatment for Alzheimer's disease.
Pre-assignment Details: Patients were excluded when in advanced or terminal stage of the disease, lived in nursing homes and when it was not possible to contact the patient.
Groups:
- Pharmacotherapy Follow-up: All the patients received pharmacotherapy workup at baseline and after the intervention.
Period: Overall Study
Arm/Group | Pharmacotherapy Follow-up
Started | 163
Completed | 55
Not Completed | 108

BASELINE CHARACTERISTICS:
Groups:
- Treatment: patients in treatment for Alzheimer's disease.
Arm/Group | Treatment
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Mini-mental State Examination (MMEE)
Description: MMEE : scale 0-30 ( ≥25 - normal aging; 21-24 - initial stage; 20-10 - middle stage; ≤9 - final stage)
Time Frame: six months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Pharmacotherapy Follow-up
Number analyzed (Participants) | 55
score
  Before | 12 (7.3)
  After | 12 (7.8)
Statistical Analysis 1: Comparison: Pharmacotherapy Follow-up; Test type: Superiority or Other; p = 0.23, t-test, 1 sided

2. Primary Outcome: Clinical Dementia Rating (CDR)
Description: CDR: scale 1-3 (0-0.5: normal aging; 1- initial stage; 2- middle stage; 3- final stage)
Time Frame: six months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Pharmacotherapy Follow-up
Number analyzed (Participants) | 55
score
  Before | 1.6 (0.08)
  After | 1.7 (0.08)
Statistical Analysis 1: Comparison: Pharmacotherapy Follow-up; Test type: Superiority or Other; p = 0.05, t-test, 1 sided

3. Secondary Outcome: Systolic Blood Pressure
Description: Systolic pressure <140 mmHg
Time Frame: weekly
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pharmacotherapy Follow-up
Number analyzed (Participants) | 55
mmHg
  Before | 136.6 (22.3)
  After | 126.7 (18.5)
Statistical Analysis 1: Comparison: Pharmacotherapy Follow-up; Test type: Superiority or Other; p = 0.03, t-test, 1 sided

4. Secondary Outcome: Total Cholesterol
Description: Total Cholesterol <200 mg/dL
Time Frame: Total Cholesterol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pharmacotherapy Follow-up
Number analyzed (Participants) | 55
mg/dL
  Before | 202.2 (41.6)
  After | 187.6 (39.5)
Statistical Analysis 1: Comparison: Pharmacotherapy Follow-up; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

5. Secondary Outcome: Triglycerides
Description: Normal level: 150mg/dL
Time Frame: three months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pharmacotherapy Follow-up
Number analyzed (Participants) | 55
mg/dL
  Before | 154.1 (63.2)
  After | 137.8 (48.7)
Statistical Analysis 1: Comparison: Pharmacotherapy Follow-up; Test type: Superiority or Other; p = 0.025, t-test, 1 sided

6. Secondary Outcome: Glycemia
Description: Normal levels: 70-99mg/dL; diabetic: >121mg/dL.
Time Frame: two months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pharmacotherapy Follow-up
Number analyzed (Participants) | 55
mg/dL
  Before | 121.9 (57.3)
  After | 93.9 (15.3)
Statistical Analysis 1: Comparison: Pharmacotherapy Follow-up; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

7. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic pressure <90 mmHg
Time Frame: weekly
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pharmacotherapy Follow-up
Number analyzed (Participants) | 55
mmHg
  Before | 75.49 (12)
  After | 73.03 (9.8)
Statistical Analysis 1: Comparison: Pharmacotherapy Follow-up; Test type: Superiority or Other; p = 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Do not apply.
Description: Do not apply.
Groups:
- Treatment: Do not apply.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No